CLINICAL TRIAL: NCT00688389
Title: Follow-up the Health Condition , Investigation of the Immuno-regulation , and the Study for Interaction of Viral Hepatitis--- Among Patients With or After Dengue Fever Infection
Brief Title: Investigation of the Immuno-regulation and Viral Hepatitis Among Patients With or After Dengue Fever Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-960195_1; CB9615
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Dengue Fever
Keywords: Dengue fever, CLEC5A, Mannose receptor, DC-SIGN, NALP,; decoy receptor 3 (DcR3), Toll-like receptors(TLRs),; (Nod)-like receptors (NLRs)
MeSH Terms: conditions — Dengue | interventions — Case-Control Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- healthy
  Interventions: Other: case/control
- DF
  Interventions: Other: case/control
- DHF
  Interventions: Other: case/control

INTERVENTIONS:
Other: case/control — case: infected dengue fever people control:healthy people

SUMMARY:
The study will collect the blood samples from 350 healthy persons and 350 persons infected with dengue fever.

DETAILED DESCRIPTION:
Research has showed that CLEC5A interacts with dengue virion directly, and is responsible for dengue virus (DV)-induced DAP12 phosphorylation. Data suggests that CLEC5A is a potential therapeutic target for dengue hemorrhagic fever (DHF)/dengue shock syndrome (DSS). This project will study the genes of CLEC5A, Mannose receptor, DC-SIGN, NALP, decoy receptor 3 (DcR3), Toll-like receptors(TLRs), and (Nod)-like receptors (NLRs) for both DF and DHF groups. In addition, serum level of decoy receptor 3 (DcR3) will be tested. The study will collect the blood samples from 350 healthy persons and 350 persons infected with dengue fever.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Dengue fever

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The samples are obtained from the Kaohsiung Medical University Chung-Ho Memorial Hospital in Kaohsiung, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2007-07; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
檢查肝臟、腎臟及其他生化功能，並分析宿主免疫調控及血小板變化機致 | 2007/7/1
  抽血20 c.c 檢查肝臟、腎臟及其他生化功能，並分析宿主免疫調控及血小板變化機致

CONTACTS AND LOCATIONS:
Locations (1):
- Kaoshing Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan